CLINICAL TRIAL: NCT04790682
Title: LIquid Biopsy to prEdict Responses To First-line immunotherapY in Metastatic Non-small Cell LUNG Cancer
Brief Title: LIquid Biopsy to prEdict Responses To First-line immunotherapY in Metastatic Non-small Cell LUNG Cancer. LIBERTY LUNG
Acronym: LIBERTYLUNG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Curie (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IC 2020-02
Record Dates: First submitted 2021-03-05; First posted 2021-03-10 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Lung Cancer
Keywords: Lung Cancer NSCLC; metastatic stage; first-line treatment with immunotherapy
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NSCLC patient in a metastatic stage eligible for 1st-line TT with immune checkpoint inhibitor. (Experimental): Patient with histologically proven Non Small Cell Lung Cancer in a metastatic stage, treatment naïve and eligible for first-line treatment with immune checkpoint inhibitor. Combination with chemotherapy is possible.
  Presence of a mutation after NGS analysis is required for ctDNA follow-up.
  Interventions: Biological: assessment of the predictive value of ctDNA level of the prominent mutant allele variation between baseline and week 6, on response to treatment according to RECIST 1.1 criteria.

INTERVENTIONS:
Biological: assessment of the predictive value of ctDNA level of the prominent mutant allele variation between baseline and week 6, on response to treatment according to RECIST 1.1 criteria. — * At pre-screening NGS analysis on tumor tissue (slides). Only patients with at least 1 mutation at NGS on the tumor tissue will ultimately be enrolled in the main study, to have the possibility to follow the mutation using ctDNA.
  * Main study will be initiated after results of the NGS and before initiation of pembrolizumab. Blood specimens will be taken with EDTA tubes or streck tubes at the time of puncture for pembrolizumab infusion at baseline before starting treatment, at 3 weeks, 6 weeks and then every 6 weeks (30 ml at Baseline then 20 ml of blood). Blood immunomonitoring will be done before starting the treatment, at 6 weeks and at 18 Week. An additional measurement will be performed if treatment is stopped before the end of the study (18 ml of blood).
  * Optional blood samples will be realized to analyse the degree of activity of the plasmatic lymphocytes before starting the treatment and at 6 weeks and (18 ml of blood).

SUMMARY:
Patient with histologically proven NSCLC in a metastatic stage, treatment naïve and eligible for first-line treatment with immune checkpoint inhibitor. Combination with chemotherapy is possible. Presence of a mutation after NGS analysis is required for ctDNA follow-up.

DETAILED DESCRIPTION:
A pre-screening consent will be obtained for NGS analysis on tumor tissue. Only patients with at least 1 mutation at NGS on the tumor tissue will ultimately be enrolled in the study, to have the possibility to follow the mutation using ctDNA. Main consent will be obtained after results of the NGS and before initiation of pembrolizumab. Computed Tomography (CT)-scan imaging will be done every 9 weeks as part of routine care practice. Blood specimens will be taken with EDTA tubes or streck tubes at the time of puncture for pembrolizumab infusion at baseline before starting treatment, at 3 weeks, 6 weeks and then every 6 weeks. Blood immunomonitoring will be done before starting the treatment, at 6 weeks and at 18 week. An additional measurement will be performed if treatment is stopped before the end of the study.

- Optional blood samples will be realized to analyse the degree of activity of the plasmatic lymphocytes.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically-proven NSCLC.
2. Age ≥ 18 years.
3. Advanced or metastatic stage IV.
4. Treatment-naïve patient.
5. Eligibility to first-line treatment with immune checkpoint inhibitor.
6. Measurable disease according to RECIST 1.1 criteria on CT-Scan.
7. Availability of expression of PD-L1 at immunohistochemistry analysis of the tumor biopsy.
8. No ALK or EGFR gene alteration.
9. Availability of tumor tissue for NGS analysis (7 slides).
10. PS 0 or 1.
11. Signed informed consent of the patient.

Exclusion Criteria:

1. No social security affiliation.
2. Person under legal protection.
3. Pregnant and breastfeeding women.

Patients can participate to another clinical trial that is not modifying immunotherapy or immunotherapy/chemotherapy treatment nor study follow-up ; after investigator's information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-05-22 (Actual); Primary Completion 2029-06-03 (Estimated); Study Completion 2030-06-03 (Estimated)

PRIMARY OUTCOMES:
ctDNA variation of the prominent mutant allele variation | 6 weeks on response to treatment defined as the proportion of patients who will achieve a complete or partial response at CT-scan based on RECIST 1.1 criteria
  ctDNA variation of the prominent mutant allele variation between baseline and week 6, on response to treatment defined as the proportion of patients who will achieve a complete or partial response at CT-scan based on RECIST 1.1 criteria.

SECONDARY OUTCOMES:
ctDNA variation of the prominent mutant allele variation | 6 weeks on response to treatment defined as the proportion of patients who will achieve a complete or partial response at CT-scan based on iRECIST criteria.
  ctDNA variation of the prominent mutant allele variation between baseline and week 6, on response to treatment defined as the proportion of patients who will achieve a complete or partial response at CT-scan based on iRECIST criteria.
Free survival | End of study
  Progression-free survival according to immune cell levels in the blood
Overall survival | End of study
  Overall survival according to immune cell levels in the blood
Survival (FS) | End of study
  Progression-free survival according to immune cell levels variations in the blood
Survival (OS) | End of study
  Overall survival according to immune cell levels variations in the blood
Progression-free | End of study
  Progression-free survival according to ctDNA level variations.
Survival | End of study
  Overall survival according to ctDNA level variations.
Response rate to the second line of treatment | End of study
  Response rate to the second line of treatment based on RECIST 1.1 and iRECIST criteria according to ctDNA level at week 6 of the second line of treatment.
Adverse events of special interest | End of study
  Adverse events of special interest of grade 3 or more (CTCAE v5.0).

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas GIRARD, PR, Study Director — INSTITUT CURIE - Medical Oncology; Pierre FUMOLEAU, Study Chair — INSTITUT CURIE - Medical Oncology
Locations (3):
- France (3):
  - Hopital Ambroise Pare, Boulogne-Billancourt
  - Institut Curie, Paris
  - Institut Curie, Saint-Cloud

IPD SHARING:
Plan to Share IPD: Yes
Sponsor will share de-identified data sets. Documents generated under the project will be disseminated in accordance with Institut Curie policies.
Supporting Information: Study Protocol, SAP
Time Frame: Data requests can be submitted starting 9 months after last article publication and will be made accessible for up to 12 months.
Access Criteria: Access to trial individual participant data can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a data sharing agreement (DSA).